CLINICAL TRIAL: NCT00808561
Title: Prospective Randomized Trial of Fistula vs. Forearm AV Graft in Patients With Poor Venous Access; Protocol #3, Version 1
Brief Title: Randomized Fistula Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment due to multiple screen failures
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol #3, V1, Fistula
Record Dates: First submitted 2008-12-12; First posted 2008-12-16 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Alternative Fistula (Active Comparator)
  Interventions: Other: Group 1: Alternative Fistula
- 2 Forearm AV Graft (Active Comparator)
  Interventions: Other: Group 2: Forearm AV Graft

INTERVENTIONS:
Other: Group 1: Alternative Fistula — Performing other autogenous AV fistulas which include various options such as brachiocephalic AV fistula, basilic or brachial vein transpositions or a variety of other strategies to maintain a primary access. The advantage would be to maintain an autogenous all venous access with less risk of infection and thrombosis.
  Arms: 1 Alternative Fistula
Other: Group 2: Forearm AV Graft — a) ePTFE (polytetrafluoroethylene) bridge AV graft typically anastomosed in the proximal forearm to the radial or brachial artery and to an antecubital vein. The advantages include a quick maturation of 2-3 weeks, excellent flow rates and high technical success rates. Although secondary patency rates approach 80% at one year postoperatively, disadvantages include a more involved surgical procedure, a lower primary patency than a well functioning AV fistula, and higher revision and infection rates.4, 5
  Arms: 2 Forearm AV Graft

SUMMARY:
The primary objective of this study is to compare two treatment strategies for establishing dialysis access in patients with unsuitable forearm veins for the standard forearm primary radio-cephalic arteriovenous fistula also known as the Brescia-Cimino fistula.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE:

Among patients with end stage renal disease (ESRD) who require hemodialysis, the maintenance of an adequate vascular access is of critical importance. As the overall population in the U.S. ages, every year a greater number of patients are being maintained on hemodialysis with an estimated Medicare expenditure in excess of 1.25 billion dollars per year.1 The complications related to dialysis access are a major determinant of patient outcomes, including morbidity and mortality, and between 16-25% of hospital admissions for dialysis patients in the U.S. are related to dialysis access complications with an estimated cost of 100 million dollars.2

For patients with ESRD requiring chronic hemodialysis, the autogenous Brescia-Cimino fistula is the consensus best choice for the creation of an AV access site for hemodialysis. This type of primary fistula uses the radial artery at the wrist and a suitable cephalic vein at the level of the wrist. The fistula typically matures in 6-8 weeks when the vein and artery are normal, and provides good flow rates with a minimal incidence of ischemia of the hand. Infection rates are extremely low and long term patency is excellent. The disadvantage is a low maturation rate when the vein has segments of fibrosis from previous IV sites or venipunctures which are common in the cephalic vein at the wrist. Difficulty with fistula maturation can lead to prolonged time with a tunneled dialysis catheter (TDC) while the patient undergoes a variety of procedures to correct the fistula and allow it to mature. Up to 40% of forearm primary Brescia-Cimino fistulas either fail to mature or occlude prior to use, and the incidence of failure of forearm fistulas is significantly higher in women compared to men. Infection rates with tunneled dialysis catheters are roughly 10 times that of fistulas or grafts; therefore, months or even years with TDCs, while fistulas mature, can have consequences. Infections are estimated to account for 14% of deaths in ESRD patients.3

In the absence of a suitable cephalic vein at the wrist or in case of poor maturation, the two main options exist. They are both acceptable in clinical practice and are chosen based on the particular clinical scenario and, to some extent, surgeon preference. The options include:

1. ePTFE (polytetrafluoroethylene) bridge AV graft typically anastomosed in the proximal forearm to the radial or brachial artery and to an antecubital vein. The advantages include a quick maturation of 2-3 weeks, excellent flow rates and high technical success rates. Although secondary patency rates approach 80% at one year postoperatively, disadvantages include a more involved surgical procedure, a lower primary patency than a well functioning AV fistula, and higher revision and infection rates.4, 5
2. Performing other autogenous AV fistulas which include various options such as brachiocephalic AV fistula, basilic or brachial vein transpositions or a variety of other strategies to maintain a primary access. The advantage would be to maintain an autogenous all venous access with less risk of infection and thrombosis. Some of these procedures, however, may involve an extensive dissection, a longer time for maturation, and the resulting fistula can be more difficult to use even if functioning well. Several procedures are also performed on occasion to aid in maturation before an AV fistula is actually available for access. In addition, a "steal" phenomenon is more common with proximal fistulas as the flow rates can be excessively high with low central resistance in the larger veins, leading to a decrease in blood flow to the hand. All of these factors often translate into prolonged central venous catheter placement (TDC) for dialysis, which has been associated with a high incidence of infection and central vein stenosis, or thrombosis.6

Because of the superior patency of primary fistulas, the Kidney Disease Outcomes Quality Initiative (K/DOQI) and the Fistula First initiative have articulated the advantages of fistulas vs. ePTFE bridge grafts for long-term dialysis access and recommended that at least 50% of patients in any region be on dialysis through a primary fistula.7 In addition, in 2006 K/DOQI set a target of 66% for prevalent fistulas by 2009.8 Many surgeons have also adopted a 100% autogenous policy because of these recommendations without a critical assessment of the potential downside of that policy.9 Others continue to use ePTFE preferentially when a cephalic vein is not available.

Although there is no doubt that in suitable patients a primary fistula is better than a prosthetic graft, there are no data to guide the best treatment strategy in the absence of a suitable forearm cephalic vein. Although K/DOQI encourages creation of primary fistulas, the multiple procedures required for fistula maturation and prolonged time with tunneled dialysis catheters, their complications may outweigh the complications of ePTFE grafts.10

ELIGIBILITY:
Inclusion Criteria:

To participate in this study, the subject MUST have all of the following for inclusion in the study:

* The subject must be > 18 years of age, male or female
* Subject requires creation of dialysis access secondary to ESRD in the opinion of the referring nephrologist
* Target arm may have a failed radiocephalic fistula
* Contralateral failed or failing access may exist
* The subject must sign a written informed consent, prior to the procedure, using a form that is approved by the local Institutional Review Board.

Exclusion Criteria:

To participate in this study, the subject may NOT HAVE any of the following at enrollment to the study:

* Target arm has existing forearm AV graft, either functional or non-functional
* Target arm has existing fistula, either functional or non-functional, other than a radio-cephalic at the wrist
* Target arm has documented subclavian vein occlusion
* Target arm has obviously suitable cephalic vein and radial artery for a primary radiocephalic fistula
* Target arm has no superficial veins existing as options for primary access. If so, a second surgeon will review the ultrasound to confirm
* Active local or systemic infection at the time of surgery
* Known hypercoagulable state (e.g., antithrombin III deficiency, antiphospholipid or anticardiolipin antibodies, Factor IV Leiden, circulating lupus anticoagulant, history of heparin-induced thrombocytopenia, Protein C or S deficiency, prothrombin mutation or a history of recurrent deep venous thrombosis and/or pulmonary embolism)
* Disseminated malignancy or other terminal condition where subject is expected to live less than 6 months.
* Previous randomization in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-12; Primary Completion 2011-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the rate of composite adverse events at one year with follow-up to 3 years. Data will be tabulated every 6 months. | 12 months

SECONDARY OUTCOMES:
Secondary endpoints: Primary, assisted primary, and secondary patency at 1 and 3 years | 3 years
Death due to access-related illness | 3 years
Death due to any cause | 3 Years
New central venous stenosis or occlusion | 3 years
Steal syndrome | 3 years
Neuropathy | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Navyash Gupta, MD, Principal Investigator — University of Pittsburgh Physicians
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States